CLINICAL TRIAL: NCT00788580
Title: S0718: Phase I Study Evaluating The Combination of GW786034 (Pazopanib; NSC-737754; IND-XXXX) and CCI-779 (Temsirolimus; NSC-683864; IND-XXXX) in Patients With Advanced Solid Tumors
Brief Title: S0718 Pazopanib and Temsirolimus in Treating Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was discontinued.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: S0718; SWOG-S0718
Record Dates: First submitted 2008-11-08; First posted 2008-11-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — temsirolimus; Immunoenzyme Techniques

INTERVENTIONS:
Drug: pazopanib hydrochloride
Drug: temsirolimus
Procedure: immunoenzyme technique
Procedure: laboratory biomarker analysis
Procedure: pharmacological study

SUMMARY:
RATIONALE: Pazopanib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Pazopanib may also blocking blood flow to the tumor. Giving pazopanib together with temsirolimus may be an effective treatment for advanced solid tumors.

PURPOSE: This phase I trial is studying the side effects and best dose of temsirolimus when given together with pazopanib in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the safety and feasibility of temsirolimus and pazopanib when given in combination in patients with advanced solid tumors.
* To recommend the maximum tolerated dose of this regimen in these patients.
* To investigate the pharmacokinetics of temsirolimus alone and in combination with pazopanib in these patients.
* To investigate the effects of this regimen on relevant biological markers.
* To preliminarily report objective response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive temsirolimus IV over 30 minutes on days 1, 8,15, and 22 and oral pazopanib hydrochloride once daily on days 4-28 in course 1 and days 1-28 in all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained periodically for evaluation of the pharmacokinetics of temsirolimus and pazopanib, plasma and serum angiogenic and cachectic factors (e.g., VEGF, bFGF, PlGF and SDF-1) by enzyme-linked immunosorbent assay, and biological markers in the mTOR/PI3/Akt, Ras/MAPK, VEGFR, PDGFR, and HIF-1 pathways.

After completion of study therapy, patients are followed for 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or pathologically verified cancer that is of advanced stage and for which there is no effective therapy

  * No lymphoma
* Measurable or nonmeasurable disease
* Previously irradiated (whole brain or gamma knife) brain metastases allowed provided there is no requirement for corticosteroids or anticonvulsants

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL (without transfusions)
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN if liver metastases present)
* Bilirubin normal
* Serum creatinine ≤ 1.5 times ULN OR measured creatinine clearance OR calculated creatinine clearance ≥ 60 mL/min
* QTC interval < 480 msec on baseline ECG OR average QTC < 480 msec on baseline plus 2 additional screening ECG's
* Fasting cholesterol < 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* No uncontrolled hypertension, arterial thrombotic event, or bleeding on therapeutic anticoagulation with warfarin or heparin (including low molecular weight heparin) within the past 6 months
* Able to swallow enteral medications
* No feeding tubes
* No intractable nausea or vomiting
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn, ulcerative colitis)
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to rapamycin analogs (e.g., sirolimus and everolimus)
* No known HIV positivity
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or serious active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Serious cardiac arrhythmia
  * History of myocardial infarction
  * Cerebrovascular accident within 3 months of study entry
  * Uncontrolled diarrhea
  * Psychiatric illness or social situation that would limit compliance with study requirements
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception, including barrier methods
* Willing to undergo pharmacokinetic (PK) sampling and blood submission for PK and translational medicine studies

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior pazopanib hydrochloride or temsirolimus
* More than 28 days since prior major surgery, chemotherapy, biologic therapy, or immunotherapy
* More than 28 days since prior investigational agents
* At least 14 days since prior radiotherapy
* No concurrent rapamycin (sirolimus)
* No concurrent enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital), CYP3A4 inducers (e.g., rifampin or St. John's wort), or CYP3A4 inhibiting agents or substrates (e.g., ketoconazole, diltiazem, or verapamil)
* No concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other type of therapy for treatment of this cancer while on this protocol

  * No live vaccines
  * Luteinizing-hormone releasing-hormone agonists allowed
* Concurrent prophylactic warfarin (≤ 1 mg/day) allowed
* Concurrent bisphosphonate or erythropoietin or its analogue allowed, if deemed appropriate by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by NCI CTCAE v3.0
Feasibility of the drug combination
Maximum tolerated dose of temsirolimus in combination with pazopanib

SECONDARY OUTCOMES:
Pharmacokinetics of temsirolimus alone and in combination with pazopanib
Relevant biological markers
Objective response as assessed by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Claire F. Verschraegen, MD, Principal Investigator — University of New Mexico Cancer Center